CLINICAL TRIAL: NCT02148237
Title: Intervention to Increase Breastfeeding Duration Among Puerto Rican Mothers
Brief Title: Increase Breastfeeding Duration Among Puerto Rican Mothers
Acronym: BFCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03HD077057 (NIH); 1R03HD077057-01A1 (NIH)
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Breastfeeding
Keywords: Breastfeeding duration; Puerto Rican mothers; WIC program; Home-based individual breastfeeding consultation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants in Treatment as Usual (TAU) will receive standard breastfeeding (BF) services from the WIC program and participate in research assessments. Standard services include an on-site and home-visiting lactation consultant, occasional one-on-one peer counseling, and an enhanced food package for BF women.
- Contingency Management (Experimental): These participants will receive usual WIC care. The frequency, duration, content, and size of the meetings and participation requirements will be the same as for the TAU group, except that this group will also receive contingency management (CM). Members will demonstrate breastfeeding and receive cash incentives weekly if they breastfeed.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Participants in this condition will receive usual WIC care in addition to Contingency Management (CM). BF will be determined by direct observation.
  Arms: Contingency Management

SUMMARY:
This study is to determine preliminary effects of home-based individual breastfeeding consultation with and without cash incentives to increase breastfeeding (BF) duration among low-income Puerto Rican mothers enrolled in a Special Supplemental Nutrition Program for Women, Infants, and Children (WIC).

DETAILED DESCRIPTION:
This study is to determine feasibility, acceptability, and preliminary effect sizes of home-based individual breastfeeding consultation alone and combined with financial incentives to increase breastfeeding (BF) duration among low-income Puerto Rican mothers. These interventions will be tested in a Women, Infants, and Children (WIC) program, which capitalizes on the current goals of WIC and on the current practice of using incentives to support BF - factors that are likely to increase potential for sustainability and dissemination of the intervention. We will follow a three phase strategy. During the Formative Phase we will consult WIC staff, Puerto Rican postpartum mothers, and experts in BF, behavioral health incentives, and WIC populations and settings to develop intervention and research manuals. During the Implementation Phase, we will pilot the interventions and research procedures. We will randomly assign 60 Puerto Rican women who initiate BF to: Treatment-as-Usual (TAU) or TAU with financial incentives (also known as Contingency Management; (CM). A bilingual breastfeeding counselor visits participants at home for problem solving issues around breastfeeding. Participants also receiving CM will receive cash incentives if they show breastfeeding. We will conduct assessments at baseline, 1, 3, and 6 months postpartum, measuring BF duration, BF exclusivity, BF self-efficacy, and infant weight gain. In the Evaluative Phase, we will examine monthly recruitment, consent, and enrollment rates, as well as attendance and retention rates for the interventions and for research participation (i.e., feasibility and acceptability).

ELIGIBILITY:
Inclusion Criteria:

1. Identify as Puerto Rican or of Puerto Rican descent
2. be able to read Spanish or English
3. currently live in the area and plan to stay until 12 months postpartum
4. be able to participate in Spanish-speaking peer-support group meetings
5. consent to participate
6. pass an informed consent quiz
7. successfully initiate BF
8. be within 15-44 years of age

Exclusion Criteria:

1. Have ongoing illicit drug use
2. have current active suicidal thoughts or a past suicide attempt, or a psychiatric hospitalization within the last 3 months
3. have untreated HIV (BF contraindicated)
4. are currently prescribed psychotropic medication (i.e., antidepressants, antipsychotics, mood stabilizers, anxiolytics)
5. have serious postpartum medical problems (e.g., postpartum hemorrhage, infections and serious jaundice requiring exchange transfusion)

Ages: 15 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Duration of breastfeeding | 6-month postpartum
  Observe breastfeeding (BF) behavior looking for one of the following indicators of successful BF in the infant: audible swallowing, a regular suck/swallow/breathe pattern, or visible milk in the infant's mouth after they are not latched anymore. For a mother who pumps milk, observation of pumping combined with observation of the resulting milk being fed to the infant will be observed.

SECONDARY OUTCOMES:
Infant weight | 1-month, 3-month, and 6-month postpartum
  An infant will be weighed at each assessment time point using a portable Health O Meter Infant Scale.

OTHER OUTCOMES:
Coercion assessment | Weekly group meetings, assessments after delivery, 1-month postpartum, 3-month postpartum, and 6-month postpartum
  The Coercion Assessment Scale (CAS) is a 11-item questionnaire that measures perceived coercion to participate in research. The items examine pressures emanating from WIC staff and the research assistant. An initial support for the instrument's internal consistency, factor structure, and discriminative validity has been provided.
Postnatal Depression | After delivery, 1-month, 3-month, and 6-month postpartum
  Edinburgh postnatal depression scale (EPDS) is a 10-item questionnaire that identifies patients at risk for perinatal depression. The EPDS was found to be sensitive and specific, especially sensitive to change in the severity of depression over time. The scale can be completed in about 5 minutes and scoring is very simple.
Breastfeeding self-efficacy scale | After delivery, 1-month, 3-month, and 6-month postpartum
  Breastfeeding self-efficacy scale (BSES) is a 39-item questionnaire to measure maternal confidence in new BF mothers. The scale has demonstrated its predictive validity showing a positive correlation between BSES scores and infant feeding patterns at 6-week postpartum. The scale has been also useful to identify new mothers with low BF confidence at high risk for premature weaning. The scale has been translated into Spanish and replicated its validity and reliability with Puerto Rican mothers.
Satisfaction survey | 6-month postpartum
  This is a brief 10-item inventory to assess the acceptability and satisfaction with the intervention It will be conducted with the 20 participants in the CM condition.. The questionnaire will include an item that (if applicable) asks why the participant did not complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yukiko Washio, Ph.D., Principal Investigator — Treatment Research Institute
Locations (1):
- Special Supplemental Nutrition Program for Women, Infants, and Children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided